CLINICAL TRIAL: NCT05573984
Title: A Natural History and Outcome Measure Discovery Study of PRPF31 Mutation-Associated Retinal Dystrophy
Brief Title: Natural History of PRPF31 Mutation-Associated Retinal Dystrophy
Status: Active, not recruiting | Type: Observational
Sponsor: PYC Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: VP001-CL001
Record Dates: First submitted 2022-09-08; First posted 2022-10-10 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Retinitis Pigmentosa; Eye Diseases, Hereditary; Retinal Dystrophies; Retinal Dystrophy Rod; Retinal Dystrophy Rod Progressive
Keywords: Retinitis Pigmentosa; Retinitis Pigmentosa Type 11; RP11; PRPF31; Retinal Dystrophy; PRPF31 Mutation-Associated Retinal Dystrophy
MeSH Terms: conditions — Retinitis Pigmentosa; Eye Diseases, Hereditary; Retinal Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Vision Cohort 1: Score of ≥ 54 ETDRS letters read and a VF diameter ≥ 10 degrees in every meridian of the central field
- Vision Cohort 2: Score of ≥ 35 ETDRS letters read and a VF diameter < 10 degrees in any meridian of the central field
- Vision Cohort 3: Score of < 35 ETDRS letters read

SUMMARY:
The purpose of this study is to characterize the natural history through temporal systemic evaluation of subjects identified with PRPF31 mutation-associated retinal dystrophy, also called retinitis pigmentosa type 11, or RP11.

Assessments will be completed to measure and evaluate structural and functional visual changes including those impacting patient quality of life associated with this inherited retinal condition and observing how these changes evolve over time.

DETAILED DESCRIPTION:
This is a multi-center, longitudinal, prospective observational natural history study of participants with a molecularly confirmed mutation in PRPF31. Approximately 50 participants (100 eyes) at approximately 5 sites will be enrolled into a uniform protocol for follow-up and evaluations. Each participant's medical record will be reviewed for historical information, and clinical data will be recorded in a secure database. Natural history data will be collected prospectively and will include ophthalmic exams, imaging studies, electrophysiological testing, functional mobility evaluations, and questionnaires. Assessments will be conducted in a standardized protocol every 16 weeks ± 4 weeks for the first year and then every 24 weeks ± 4 weeks for up to approximately 4 years after each participant's baseline visit (Visit 2).

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following in order to be enrolled into the study:

1. Male or female, ≥ 10 years of age at baseline (Visit 2).
2. Have a clinical and molecular diagnosis of PRPF31 mutation-associated retinal dystrophy.
3. If ≥ 18 years of age, understand the language of the informed consent and are willing and able to provide written informed consent prior to any study procedures. If < 18 years of age, are willing to assent to study participation in writing and have a legally authorized representative provide written informed consent on your behalf.
4. Are willing to comply with the instructions and attend all scheduled study visits.

Exclusion Criteria:

Participants or, in the case of ocular-specific criteria, individual eyes with any of the following will not be allowed to participate in this study:

1. Have any uncontrolled systemic disease that, in the opinion of the Investigator, would preclude participation in the study (e.g., infection, uncontrolled elevated blood pressure, cardiovascular disease, or glycemic control issues) or put the participant at risk due to study procedures.
2. Have mutations in genes that cause autosomal dominant retinitis pigmentosa (adRP), X-linked retinitis pigmentosa (XLRP), or presence of biallelic mutations in autosomal recessive RP/retinal dystrophy genes other than PRPF31 mutations.
3. Have used anti-vascular endothelial growth factor (VEGF) agents or corticosteroid injections or implants.
4. Have had Ozurdex® implants placed within 3 months or Retisert® or Iluvien® implants placed within 3 years prior to Visit 2.
5. Within 3 months prior to Visit 2, have undergone any vitreoretinal surgery (scleral buckle, pars plana vitrectomy, retrieval of a dropped nucleus or intraocular lens, radial optic neurotomy, sheathotomy, cyclodestructive procedures or multiple filtration surgeries [2 or more], etc.) or any other ocular surgery.
6. Have ocular media opacity or poor pupillary dilation that prohibits quality ophthalmic evaluation or photography.
7. Have used any investigational drug or device within 90 days or 5 estimated half-lives of Visit 2, whichever is longer, or plan to participate in another study of drug or device during the study period.
8. Have received any prior cell or gene therapy for a retinal condition.
9. Have a history of illicit drug use or alcohol dependency.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of approximately 50 participants (100 eyes) with a genetically confirmed PRPF31 mutation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Best Corrected Visual Acuity (BCVA) | Baseline through Year 4
  BCVA letter score utilizing ETDRS (Early Treatment Diabetic Retinopathy Study) or BRVT (Berkeley Rudimentary Vision Test) for patients not able to see letters
Change in Best Corrected Low Luminance Visual Acuity (LLVA) | Baseline through Year 4
  Best corrected LLVA letter score measured using the ETDRS charts and a special light filter lens
Change from Baseline in Retinal Thickness | Baseline through Year 4
  Retinal thickness is measured using spectral domain optical coherence tomography (SD-OCT), as measured by the central reading center
Change from Baseline in Ellipsoid Zone (EZ) Area | Baseline through Year 4
  Change in EZ area measured using spectral domain optical coherence tomography (SD-OCT), as measured by the central reading center
Change from Baseline in Ellipsoid Zone (EZ) Volume | Baseline through Year 4
  Change in EZ volume measured using spectral domain optical coherence tomography (SD-OCT), as measured by the central reading center
Change from Baseline in Visual Field Sensitivity | Baseline through Year 4
  Visual field sensitivity measured by static perimetry with topographic analysis-Hill of Vision conducted by the central reading center
Change from Baseline in Mean Macular Sensitivity | Baseline through Year 4
  Mean macular sensitivity measured on guided microperimetry
Change from Baseline in Fixation Stability | Baseline through Year 4
  Fixation stability as measured by Macular Integrity Assessment (MAIA) microperimeter
Change from Baseline in Full Field Retinal Sensitivity | Baseline through Year 4
  Dark-adapted visual sensitivity via full-field stimulus threshold (FST) measurement
Change from Baseline in Electrical response | Baseline through Year 4
  Electrical response measured using Full-field electroretinogram (ERG) with specific stimuli
Characterization of Changes of the Retina with Fundus Photography | Baseline through Year 4
  Abnormalities captured by fundus photography
Change from Baseline in Area of Fundus Autofluorescence (FAF) | Baseline through Year 4
  Area of hypo-autofluorescence captured by fundus autofluorescence (FAF)
Change from Baseline in Functional Vision | 3 times prior to Month 4
  Functional vision is measured with a functional mobility course (Ora-VNC™) score
Change in Patient Reported Outcome Measures using Michigan Retinal Degeneration Questionnaire (MRDQ) | Baseline through Year 4
  Responses on the MRDQ, a validated patient reported outcomes measure designed in accordance with U.S. FDA guidelines, specifically for conditions of inherited retinal degeneration (IRDs)
Change in Patient Reported Outcome Measures using Patient Global Impression of Severity (PGI-S) scale | Baseline through Year 4
  Responses on the PGI-S to assess severity of the patient's condition
Change in Patient Reported Outcome Measures using Patient Global Impression of Change (PGI-C) scale | Baseline through Year 4
  Responses on the PGI-C to assess change of the patient's condition
Genomic Analysis for Study Eligibility | Screening
  Whole exome genomic analysis
Ocular Adverse Events (AEs) | Screening through Year 4
  Frequency of ocular adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Sreenivasu Mudumba, PhD, Study Chair — PYC Therapeutics
Locations (7):
- United States (5):
  - University of California San Francisco, San Francisco, California
  - University of Florida Health, Jacksonville, Florida
  - University of Michigan Kellogg Eye Center, Ann Arbor, Michigan
  - Oregon Health and Science University - Casey Eye Institute, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas
- Australia (2):
  - Lions Eye Institute, Nedlands, Western Australia
  - Centre For Eye Research Australia (CERA) - Retinal Gene Therapy Unit, East Melbourne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hartong DT, Berson EL, Dryja TP. Retinitis pigmentosa. Lancet. 2006 Nov 18;368(9549):1795-809. doi: 10.1016/S0140-6736(06)69740-7. PMID 17113430
- [Background] Ferrari S, Di Iorio E, Barbaro V, Ponzin D, Sorrentino FS, Parmeggiani F. Retinitis pigmentosa: genes and disease mechanisms. Curr Genomics. 2011 Jun;12(4):238-49. doi: 10.2174/138920211795860107. PMID 22131869
- [Background] Rio Frio T, Wade NM, Ransijn A, Berson EL, Beckmann JS, Rivolta C. Premature termination codons in PRPF31 cause retinitis pigmentosa via haploinsufficiency due to nonsense-mediated mRNA decay. J Clin Invest. 2008 Apr;118(4):1519-31. doi: 10.1172/JCI34211. PMID 18317597
- [Background] Sullivan LS, Bowne SJ, Seaman CR, Blanton SH, Lewis RA, Heckenlively JR, Birch DG, Hughbanks-Wheaton D, Daiger SP. Genomic rearrangements of the PRPF31 gene account for 2.5% of autosomal dominant retinitis pigmentosa. Invest Ophthalmol Vis Sci. 2006 Oct;47(10):4579-88. doi: 10.1167/iovs.06-0440. PMID 17003455
- [Background] Venturini G, Rose AM, Shah AZ, Bhattacharya SS, Rivolta C. CNOT3 is a modifier of PRPF31 mutations in retinitis pigmentosa with incomplete penetrance. PLoS Genet. 2012;8(11):e1003040. doi: 10.1371/journal.pgen.1003040. Epub 2012 Nov 8. PMID 23144630
- [Background] Vithana EN, Abu-Safieh L, Allen MJ, Carey A, Papaioannou M, Chakarova C, Al-Maghtheh M, Ebenezer ND, Willis C, Moore AT, Bird AC, Hunt DM, Bhattacharya SS. A human homolog of yeast pre-mRNA splicing gene, PRP31, underlies autosomal dominant retinitis pigmentosa on chromosome 19q13.4 (RP11). Mol Cell. 2001 Aug;8(2):375-81. doi: 10.1016/s1097-2765(01)00305-7. PMID 11545739
- [Background] Wheway G, Douglas A, Baralle D, Guillot E. Mutation spectrum of PRPF31, genotype-phenotype correlation in retinitis pigmentosa, and opportunities for therapy. Exp Eye Res. 2020 Mar;192:107950. doi: 10.1016/j.exer.2020.107950. Epub 2020 Jan 31. PMID 32014492
- [Background] Food and Drug Administration. Rare Diseases: Natural History Studies for Drug Development. Draft Guidance for Industry 2019. https://www.fda.gov/media/122425/download